CLINICAL TRIAL: NCT03401229
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Phase 3 Efficacy and Safety Study Of Benralizumab in Patients With Severe Nasal Polyposis
Brief Title: Efficacy and Safety Study of Benralizumab for Patients With Severe Nasal Polyposis
Acronym: OSTRO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3252C00001; 2017-003675-61 (EudraCT Number); NCT03627286 (obsolete NCT alias)
Record Dates: First submitted 2017-12-13; First posted 2018-01-17 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Nasal Polyposis
Keywords: Polyps; Nasal polyps; Nasal polyposis; Nose diseases; Respiratory tract diseases; Otorhinolaryngologic diseases; Benralizumab; Mometasone furoate
MeSH Terms: conditions — Nasal Polyps; Polyps; Nose Diseases; Respiratory Tract Diseases; Otorhinolaryngologic Diseases | interventions — benralizumab; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab 30mg SC + MF (Experimental): SC - subcutaneously MF - Mometasone Furoate
  Interventions: Biological: Benralizumab 30 mg SC + Mometasone Furoate
- Placebo SC + MF (Placebo Comparator)
  Interventions: Biological: Matching placebo SC + Mometasone Furoate

INTERVENTIONS:
Biological: Benralizumab 30 mg SC + Mometasone Furoate — Benralizumab injection is 30mg/ml SC clear to opalescent, colourless to yellow solution in accessorized pre-filled syringe.
  Benralizumab 30 mg SC will be injected every 4 weeks for the first 3 doses - Weeks 0 , 4 and 8 and every 8 weeks thereafter - Weeks 16, 24, 32, 40 and 48. Total of 8 doses.
  Mometasone Furoate Nasal Spray (MFNS) - intranasal corticosteroid - 2 doses (1 dose = 50 micrograms/actuation) in each nostril twice daily. Total daily dose of 400mcg. MFNS will be used for a minimum of 4 weeks prior to randomization and will be continued throughout the study.
  Arms: Benralizumab 30mg SC + MF
Biological: Matching placebo SC + Mometasone Furoate — Matching placebo injection is SC clear to opalescent, colourless to yellow solution in accessorized pre-filled syringe.
  Matching placebo SC will be injected every 4 weeks for the first 3 doses - Weeks 0 , 4 and 8 and every 8 weeks thereafter - Weeks 16, 24, 32, 40 and 48. Total of 8 doses.
  Mometasone Furoate Nasal Spray (MFNS) - intranasal corticosteroid - 2 doses (1 dose = 50 micrograms/actuation) in each nostril twice daily. Total daily dose of 400mcg. MFNS will be used for a minimum of 4 weeks prior to randomization and will be continued throughout the study.
  Arms: Placebo SC + MF

SUMMARY:
The aim of this present study is to investigate the use of benralizumab as treatment for severe nasal polyposis. The effect of benralizumab on nasal polyps will be assessed over a 56 weeks of treatment period in patients with severe bilateral nasal polyposis who are still symptomatic despite standard of care therapy, i.e current use of intranasal corticosteroids (INCS) and prior surgery and/or use of systemic corticosteroids. The first 200 patients that complete the 56-week treatment will have a 6 month follow-up (FU) period without dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions, listed in the informed consent form (ICF) and in protocol.
2. Provision of signed and dated, written informed consent form (ICF) prior to any mandatory study specific procedures, sampling, and analyses and according to international guidelines and/or applicable European Union (EU) guidelines.
3. Provision of signed and dated written genetic informed consent in patients that agree to participate in the genetic sampling, prior to collection of sample for genetic analysis.
4. Female or male patients aged 18 to 75 years inclusive, at the time of signing the ICF.
5. Patients with bilateral sinonasal polyposis that, despite treatment with a stable dose of intranasal corticosteroids (INCS) for at least 4 weeks prior to V1, in addition to history of treatment with systemic (SCS -oral, parenteral) or prior surgery for nasal polyposis (NP), have severity consistent with a need for surgery as described by:

   * A minimum total Nasal Polyp Score (NPS) of 5 out of a maximum score of 8 (with a unilateral score of at least 2 for each nostril) at V1, and continuously maintained at V2 to meet the randomization criterion, as determined by the study Imaging Core Lab;
   * Ongoing symptoms for at least 12 weeks prior to V1;
   * Patient-reported moderate to severe nasal blockage score (NBS) 2 or 3 over the 2-weeks prior to V1 (2-week recall assessment of symptoms, scores 0-none to 3-severe).
6. SNOT-22 total score ≥ 30 at enrolment.

   Patient must meet the following criteria (points 7-10) at the randomization visit:
7. At least 8 days of evaluable daily diary data in the 14-day period prior to randomization (baseline bi-weekly mean score collected from study Day -13 to study Day 0).
8. At randomization, a bi-weekly mean NBS ≥ 1.5.
9. SNOT-22 total score ≥ 30 at randomization.
10. At least 70% compliance with INCS during the run-in period based on daily diary.
11. Patients with a minimum weight of 40kg.
12. Negative serum pregnancy test result and a negative urine pregnancy test at randomization for female patients of childbearing potential.
13. Women of childbearing potential (WOCBP) must use an effective form of birth control as defined in the Clinical Study Protocol (CSP).

15. Male subjects who are sexually active must be surgically sterile at least one year prior to Visit 1 or must use an adequate method of contraception (condom or condom with spermicide depending on local regulations) from the first dose of IP until 16 weeks after their last dose. Men with a partner or partners who is (are) not of childbearing potential are exempt of these requirements

Exclusion Criteria:

1. Patients who have undergone any nasal and/or sinus surgery within 3 months prior to V1.
2. Patients with conditions or concomitant disease that makes them non evaluable for the co-primary efficacy endpoint such as:

   * Unilateral antrochoanal polyps;
   * Nasal septal deviation that occludes at least one nostril;
   * Acute sinusitis, nasal infection, or upper respiratory infection at screening or in the 2 weeks before screening;
   * Current rhinitis medicamentosa;
   * Allergic fungal rhinosinusitis (AFRS) or Allergic fungal sinusitis (AFS);
   * Nasal cavity tumors.
3. Clinically important comorbidities that could confound interpretation of clinical efficacy results including, but not limited to: active upper or lower respiratory tract infection, cystic fibrosis, primary ciliary dyskinesia, eosinophilic diseases other than asthma (e.g. allergic bronchopulmonary aspergillosis/mycosis, eosinophilic granulomatosis with polyangitis [Churg-Strauss syndrome], hypereosinophilic syndromes), granulomatosis with polyangitis (Wegener's granulomatosis), Young's syndrome, etc.
4. Any disorder, including but not limited to: cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator or AstraZeneca and could:

   * Affect the safety of the patient throughout the study;
   * Influence the findings of the studies or their interpretations;
   * Impede the patient's ability to complete the entire duration of study.
5. Patients experiencing an asthma exacerbation requiring systemic (oral and/or parenteral) corticosteroids treatment or hospitalization (>24hrs) for treatment of asthma within 4 weeks prior to V1.
6. History of anaphylaxis to any biologic therapy or vaccine.
7. Known history of allergy or reaction to any component of the Investigational Product (IP) formulation.
8. History of Guillain-Barré syndrome.
9. A helminth parasitic infection diagnosed within 24 weeks prior to V1 and has not been treated with, or has failed to respond to standard of care therapy.
10. Current malignancy, or history of malignancy, except for: - Patients who have had basal cell carcinoma, localized squamous cell carcinoma of the skin, or in situ carcinoma of the cervix are eligible provided that patient is in remission and curative therapy was completed at least 12 months prior to V1; - Patients who have had other malignancies are eligible provided that the patient is in remission and curative therapy was completed at least 5 years prior to V1.

    NOTE: Hormonal therapy is allowed. As long as the cancer is in remission for 5 years, the patient is eligible.
11. Any clinically significant cardiac disease or any electrocardiogram (ECG) abnormality obtained during the screening/run-in period, which may put the patient at risk or interfere with study assessments.
12. Positive hepatitis B surface antigen, or hepatitis C virus antibody serology (confirmed by additional testing, e.g. hepatitis C RNA test, if indicated), or a positive medical history for hepatitis B or C (Note: Patients with history of hepatitis B vaccination without history of hepatitis B are allowed to enroll).
13. History of known immunodeficiency disorder, including a positive human immunodeficiency virus (HIV) test.
14. Infection requiring systemic antibiotics (Ab) within 14 days prior to V1
15. Use of immunosuppressive medication (including but not limited to: methotrexate, troleandomycin, cyclosporine, azathioprine, or any experimental anti-inflammatory therapy) within 3 months prior to V1.
16. Receipt of any marketed or investigational biologic products (monoclonal or polyclonal antibody) within 6 months or 5 half-lives prior to the date informed consent, is obtained, whichever is longer, prior to V1 and during the study period. This also applies to patients who previously participated in clinical studies and were treated with monoclonal antibodies (e.g. mepolizumab, reslizumab, dupilumab, omalizumab). Note that this restriction do not apply to patients, who are confirmed to have only received treatment with placebo.
17. Previous receipt of benralizumab.
18. Receipt of immunoglobulin or blood products within 30 days prior to V1.
19. Receipt of live attenuated vaccines 30 days prior to the date of randomization.
20. Receipt of any investigational drug within 30 days or 5 half-lives whichever is longer prior to randomization.
21. Receipt of systemic corticosteroid 4 weeks prior to V1, or a scheduled systemic corticosteroid treatment during the study period.

    NOTE: Sustained release steroids (e.g. Kenalog [Triamcinolone acetonide]) or depot injections require minimum 6 weeks washout prior to V1.
22. Receipt of leukotriene antagonist/modifiers for patients who were not on a continuous stable dose for ≥30 days prior to V1.
23. Concurrent enrolment in another clinical drug interventional trial.
24. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥ 3 times the upper limit of normal (ULN) confirmed during screening period.
25. Previous randomization in the present study.
26. Planned major surgical procedures or scheduled NP surgery at the time of the study enrolment and randomization.
27. Initiated or is being maintained on an aspirin desensitization regimen for the management of aspirin exacerbated respiratory disease (AERD) at the time of study enrolment or during the run-in period.
28. For women only - currently pregnant (or intend to become pregnant), breastfeeding or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bachert, Prof. dr. h.c., Principal Investigator — University Hospital Ghent, de Pintelaan 185, 9000 Ghent, Belgium
Locations (86):
- United States (40):
  - Research Site, Birmingham, Alabama
  - Research Site, Fresno, California
  - Research Site, Huntington Beach, California
  - Research Site, La Mesa, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Roseville, California
  - Research Site, Walnut Creek, California
  - Research Site, Centennial, Colorado
  - Research Site, Glenwood Springs, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Lake Mary, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Des Moines, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, Lincoln, Nebraska
  - Research Site, Hewlett, New York
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, Plainview, New York
  - Research Site, The Bronx, New York
  - Research Site, White Plains, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Conroe, Texas
  - Research Site, Houston, Texas
  - Research Site, North Logan, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Spokane, Washington
- Austria (5):
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Sankt Pölten
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
- Canada (8):
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Trois-Rivières, Quebec
- Denmark (9):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Hillerød
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Køge
  - Research Site, Næstved
  - Research Site, Odense C
  - Research Site, Vejle
- Germany (10):
  - Research Site, Aschaffenburg
  - Research Site, Berlin
  - Research Site, Dreieich
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Göttingen
  - Research Site, Heidelberg
  - Research Site, Lübeck
  - Research Site, Münster
  - Research Site, Wiesbaden
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Veszprém
- Poland (5):
  - Research Site, Lodz
  - Research Site, Nadarzyn
  - Research Site, Strzelce Opolskie
  - Research Site, Warsaw
  - Research Site, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Bachert C, Han JK, Desrosiers MY, Gevaert P, Heffler E, Hopkins C, Tversky JR, Barker P, Cohen D, Emson C, Martin UJ, Shih VH, Necander S, Kreindler JL, Jison M, Werkstrom V. Efficacy and safety of benralizumab in chronic rhinosinusitis with nasal polyps: A randomized, placebo-controlled trial. J Allergy Clin Immunol. 2022 Apr;149(4):1309-1317.e12. doi: 10.1016/j.jaci.2021.08.030. Epub 2021 Sep 29. PMID 34599979
- [Derived] Geng B, Dilley M, Anterasian C. Biologic Therapies for Allergic Rhinitis and Nasal Polyposis. Curr Allergy Asthma Rep. 2021 Jun 10;21(6):36. doi: 10.1007/s11882-021-01013-y. PMID 34110505
- See also: The redacted CSP. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3252C00001&attachmentIdentifier=2230117a-5097-441f-b83c-abd127835e60&fileName=d3252c00001-csp-v4_final_signed_Redacted.pdf&versionIdentifier=
- See also: The redacted SAP. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3252C00001&attachmentIdentifier=dac11fb4-fec1-4658-a069-6959efb08d21&fileName=d3252c00001-sap-ed-3_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 413 participants were randomized to receive treatment in study D3250C00001 (OSTRO) with benralizumab 30 mg or placebo. Of the 413 patients randomized, 410 (99.3%) received treatment with study drug. 207 (50.5%) patients received benralizumab 30 mg and 203 (49.5%) patients received placebo
Pre-assignment Details: In OSTRO, at the first visit, ie, the enrollment visit 1, patients were evaluated regarding the protocol mandated inclusion and exclusion criteria. After enrolment, eligible patients entered a 5-week screening/run in period on a stable dose of study provided Mometasone Furoate Nasal Spray (MFNS).
Groups:
- Benra 30 mg: Benra administered every 4 weeks for the first 3 doses - Weeks 0, 4 and 8 and every 8 weeks thereafter - Weeks 16, 24, 32, 40 and 48.
- Placebo: Placebo administered every 4 weeks for the first 3 doses - Weeks 0, 4 and 8 and every 8 weeks thereafter - Weeks 16, 24, 32, 40 and 48.
Period: Overall Study
Arm/Group | Benra 30 mg | Placebo
Started | 207 | 203
Completed | 167 | 166
Not Completed | 40 | 37
Not completed — Lost to Follow-up | 2 | 1
Not completed — Other | 1 | 3
Not completed — Adverse Event | 8 | 6
Not completed — Withdrawal by Subject | 29 | 26
Not completed — COVID-19 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set: All patients randomized and receiving any IP are included in the full analysis set (FAS), irrespective of their protocol adherence and continued participation in the study. Patients are analyzed according to their randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Benra 30 mg | Placebo | Total
Number analyzed (Participants) | 207 | 203 | 410
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.1 (12.38) | 50.2 (13.91) | 50.2 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 82 | 147
  Male | 142 | 121 | 263
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 197 | 190 | 387
  Black or African American | 4 | 8 | 12
  American Indian or Alaska Native | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Other | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total NPS at Week 40
Description: Change from baseline in total nasal polyps score (NPS) at week 40 was defined as the endpoint value at week 40 minus the baseline value. The total NPS was the sum of the right and left nostril scores and maximum total NPS is 8, as evaluated by nasal endoscopy and the left and right score were based on central read with scale from 0 to 4 where higher score reflects heavier bilateral nasal polyp burden. Baseline was the last valid value on or prior to the date of randomization. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied. In ANCOVA, a hybrid method of WP after NP surgery, WOCF after SCS_NP and multiple imputation (MI) assuming missing at random were used to build the complete imputation datasets for the analysis.
Time Frame: Baseline to week 40
Population: Full analysis set: All patients randomized and receiving any IP are included in the full analysis set (FAS), irrespective of their protocol adherence and continued participation in the study. Patients are analyzed according to their randomized treatment. Patients who had not been rescued and whose post-baseline observation was missing at the timepoint of interest are excluded from this analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 187 | 187
Score on a scale | -0.36 (1.66) | 0.17 (1.18)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; The primary analysis compared the changes from baseline of benralizumab with placebo. H0: The change from baseline in total NPS and/or the change from baseline in NBS are similar between benralizumab and placebo. H1: Both of the change from baseline in total NPS and the change from baseline in NBS are different between benralizumab and placebo; Test type: Superiority; p < 0.0001, ANCOVA — To account for multiplicity, a pre-specified testing strategy was followed to control the overall type I error rate. Both of the co-primary endpoints were tested at 0.01 (two-sided); ANCOVA following hybrid WP/WOCF and MI (assuming MAR), adjusting for treatment, baseline score, region (US/Non-US) and baseline comorbid asthma status; Mean Difference (Net) = -0.570, 95% CI 2-sided [-0.852 to -0.289]

2. Primary Outcome: Change From Baseline in NBS at Week 40
Description: Change from baseline in nasal blockage score (NBS) at week 40 was defined as the endpoint value at week 40 minus the baseline value. The NBS was captured by an item in NPSD. Patients were asked to rate the severity of their worst nasal blockage over the past 24 hours using the following response options: 0-none; 1-mild; 2-moderate; 3-severe. The NBS and the changes from baseline were summarized every two weeks (bi-weekly). Baseline was the average of daily responses from Day -13 to Day 1. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied. In ANCOVA, a hybrid method of the WP after NP surgery, WOCF after SCS_NP and multiple imputation (MI) assuming missing at random were used to build the complete imputation datasets for the analysis.
Time Frame: Baseline to week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 181
Score on a scale | -0.68 (1.02) | -0.41 (0.89)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0048, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.270, 95% CI 2-sided [-0.458 to -0.083]

3. Secondary Outcome: Change From Baseline in SNOT-22 at Week 40
Description: Change from baseline in SinoNasal outcome test (SNOT-22) at week 40 was defined as the endpoint value at week 40 minus the baseline value. The SNOT-22 is a condition specific health-related quality of life assessment which captures patient-reported physical problems, functional limitations, and emotional consequences of sinonasal conditions. The total score is the sum of item scores and has a range from 0 to 110 (higher scores indicate poorer outcomes). Baseline was the last valid value on or prior to the date of randomization. Data collected after NP surgery and/or SCS_NP were set to missing. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied. In ANCOVA, a hybrid method of WP after NP surgery, WOCF after SCS_NP and multiple imputation (MI) assuming missing at random were used to build the complete imputation datasets for the analysis.
Time Frame: Baseline to week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 193 | 190
Score on a scale | -15.2 (30.47) | -10.7 (31.64)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; This endpoint compared the changes from baseline of benralizumab with placebo. H0: The change from baseline in SNOT-22 total score is similar between benralizumab and placebo. H1: The change from baseline in SNOT-22 total score is different between benralizumab and placebo; Test type: Superiority; p = 0.0821, ANCOVA — Since both primary endpoints were significant at significant level of 0.01 level, this endpoint was tested at significant level of 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -5.212, 95% CI 2-sided [-11.087 to 0.664]

4. Secondary Outcome: Time to First NP Surgery and/or SCS Use for NP to Week 56
Description: The cumulative percentage and the corresponding 95% CI are based on the Kaplan-Meier estimates. Patients can have more than 1 rescue category during the study, and the first rescue per patient is considered. The time to first nasal polyposis (NP) surgery and/or systemic corticosteroids (SCS) use for NP up to week 56 was calculated based on the earliest occurrence of NP surgery and/or SCS use for NP and was calculated as follows: Time to first NP surgery and/or SCS use for NP = Earlier of (Start date of first NP surgery, Start date of first SCS use for NP) - date of randomization + 1. For patients who did not experience any surgery or SCS use for NP, the time to event was censored at earlier of (date of their week 56 visit, date of discontinuation).
Time Frame: Baseline to week 56
Population: Full analysis set: All patients randomized and receiving any IP are included in the full analysis set (FAS), irrespective of their protocol adherence and continued participation in the study. Patients are analyzed according to their randomized treatment. Number of patients analyzed is number of patients who had NP surgery and/or SCS use.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 207 | 203
months | 35.5 [29.3 to 42.5] | 46.5 [39.7 to 53.8]
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; This endpoint compared the rate of incidence of first NP surgery and/or SCS use for NP between benralizumab and placebo. H0: The rate is similar between benralizumab and placebo. H1: the rate is different between benralizumab and placebo. Hazard ratio is benralizumab vs placebo and HR less than 1 indicates longer time to event; Test type: Superiority; p = 0.0660, Regression, Cox — Based on pre-specified testing strategy, this endpoint was not tested for statistical significance and the p-value was considered nominal because test for change from baseline in SNOT-22 at week 40 was not statistically significant; A Cox proportional hazards model including covariates treatment group, region (US/Non-US) and baseline comorbid asthma status; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.55 to 1.02]

5. Secondary Outcome: Time to the First NP Surgery up to Week 56
Description: The cumulative percentage and the corresponding 95% CI are based on the Kaplan-Meier estimates. Patients can have more than 1 rescue category during the study, and the first rescue per patient is considered. The time to first nasal polyposis (NP) surgery up to week 56 was calculated based on the earliest occurrence of NP surgery and was calculated as follows: Time to first NP surgery=Start date of first NP surgery - date of randomization + 1. For patients who did not experience any surgery, the time to event was censored at earlier of (date of their week 56 visit, date of discontinuation).
Time Frame: Baseline to week 56
Population: Full analysis set: All patients randomized and receiving any IP are included in the full analysis set (FAS), irrespective of their protocol adherence and continued participation in the study. Patients are analyzed according to their randomized treatment. Number of patients analyzed is number of patients who had NP surgery.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 207 | 203
months | 16.6 [12.1 to 22.5] | 19.5 [14.5 to 25.9]
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; The endpoint compared the rate of incidence of first NP surgery between benralizumab and placebo. H0: The rate is similar between benralizumab and placebo. H1: the rate is different between benralizumab and placebo. Hazard ratio (HR) is benralizumab vs placebo and HR less than 1 indicates longer time to event; Test type: Superiority; p = 0.5008, Regression, Cox — Based on pre-specified testing strategy, this endpoint was not tested for statistical significance and the p-value was considered nominal; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.53 to 1.36]

6. Secondary Outcome: Change From Baseline in DSS at Week 40
Description: Change from baseline in difficulty with sense of smell (DSS) at week 40 was defined as the endpoint value at week 40 minus the baseline value. The DSS is captured by an item in the NPSD. Severity of worst difficulty with sense of smell over the past 24 hours was rated with response options: 0-none; 1-mild; 2-moderate; 3-severe. The DSS and the changes from baseline were summarized every two weeks (bi-weekly). Baseline was the average of daily responses from Day -13 to Day 1. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids use for NP (SCS_NP) were set to missing. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied. In ANCOVA, a hybrid method of WP after NP surgery, WOCF after SCS_NP and multiple imputation (MI) assuming missing at random were used to build the complete imputation datasets for the analysis.
Time Frame: Baseline to week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 181
Score on a scale | -0.34 (0.74) | -0.16 (0.65)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; This endpoint compared the changes from baseline DSS score of benralizumab with placebo. H0: The change from baseline in DSS score is similar between benralizumab and placebo. H1: The change from baseline in DSS score is different between benralizumab and placebo; Test type: Superiority; p = 0.0029, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.218, 95% CI 2-sided [-0.361 to -0.074]

7. Secondary Outcome: Change From Baseline in NPS at Week 56
Description: Change from baseline in total nasal polyps score (NPS) at week 56 was defined as the endpoint value at week 56 minus the baseline value. The total NPS is the sum of the right and left nostril scores, as evaluated by nasal endoscopy and the left and right score are based on central read with scale from 0 to 4 where higher score reflects heavier bilateral nasal polyp burden. Baseline was the last valid value on or prior to the date of randomization. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied. In ANCOVA, a hybrid method of WP after NP surgery, WOCF after SCS_NP and multiple imputation (MI) assuming missing at random were used to build the complete imputation datasets for the analysis.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 161 | 171
Score on a scale | -0.22 (1.76) | 0.18 (1.44)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; This endpoint compared the changes from baseline of benralizumab with placebo. H0: The change from baseline in NPS is similar between benralizumab and placebo. H1: The change from baseline in NPS is different between benralizumab and placebo; Test type: Superiority; p = 0.0054, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.475, 95% CI 2-sided [-0.810 to -0.141]

8. Secondary Outcome: Change From Baseline in NBS at Week 56
Description: Change from baseline in nasal blockage score (NBS) at week 56 was defined as the endpoint value at week 56 minus the baseline value. The NBS is captured by an item in the NPSD. Patients were asked to rate the severity of their worst nasal blockage over the past 24 hours using the following response options: 0-none; 1-mild; 2-moderate; 3-severe. The NBS and the changes from baseline were summarized every two weeks (bi-weekly). Baseline was the average of daily responses from Day -13 to Day 1. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied. In ANCOVA, a hybrid method of WP after NP surgery, WOCF after SCS_NP and multiple imputation (MI) assuming missing at random were used to build the complete imputation datasets for the analysis.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 179 | 175
Score on a scale | -0.68 (1.03) | -0.38 (0.91)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; This endpoint compared the changes from baseline of benralizumab with placebo. H0: The change from baseline in NBS is similar between benralizumab and placebo. H1: The change from baseline in NBS is different between benralizumab and placebo; Test type: Superiority; p = 0.0032, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.287, 95% CI 2-sided [-0.477 to -0.096]

9. Secondary Outcome: Change From Baseline in SNOT-22 at Week 56
Description: Change from baseline in SinoNasal outcome test (SNOT-22) at week 56 was defined as the endpoint value at week 56 minus the baseline value. The SNOT-22 is a condition specific health-related quality of life assessment which captures patient-reported physical problems, functional limitations, and emotional consequences of sinonasal conditions. The total score is range from 0 to 110 (higher scores indicate poorer outcomes). Baseline was the last valid value on or prior to the date of randomization. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied. In ANCOVA, a hybrid method of WP after NP surgery, WOCF after SCS_NP and multiple imputation (MI) assuming missing at random were used to build the complete imputation datasets for the analysis.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 190 | 184
Score on a scale | -15.1 (33.55) | -7.9 (33.22)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0188, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -7.492, 95% CI 2-sided [-13.741 to -1.243]

10. Secondary Outcome: Change From Baseline in DSS at Week 56
Description: Change from baseline in difficulty with sense of smell (DSS) at week 56 was defined as the endpoint value at week 56 minus the baseline value. The DSS is captured by an item in the NPSD with response options: 0-none; 1-mild; 2-moderate; 3-severe to rate the severity of their worst difficulty with sense of smell over past 24 hours. The DSS and the changes from baseline were summarized every two weeks (bi-weekly). Baseline was the average of daily responses from Day -13 to Day 1. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied. In ANCOVA, a hybrid method of WP after NP surgery, WOCF after SCS_NP and multiple imputation (MI) assuming missing at random were used to build the complete imputation datasets for the analysis.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 179 | 175
Score on a scale | -0.39 (0.79) | -0.21 (0.65)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0023, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.237, 95% CI 2-sided [-0.389 to -0.084]

11. Secondary Outcome: Change From Baseline in LMS at EOT/IPD
Description: Change from baseline in Computed tomography (CT) Lund Mackay Score (LMS) at end of treatment (EOT)/investigational product discontinuation (IPD) was defined as the endpoint value at EOT/IPD minus the baseline value. The LMS evaluates the patency using a 0-2 scale (0-normal; 1-partial opacification; and 2-total opacification) of each sinus (maxillary, anterior ethmoid, posterior ethmoid, sphenoid, frontal sinus on each side). The osteomeatal complex is graded as 0- not occluded or 2-occluded. The total CT score is the sum of the scores from all the sinus and ranges from 0 to 24. The minimum is 0 and higher score indicates worse outcome. The analysis used the data collected after systemic corticosteroids for nasal polyposis (SCS_NP). A composite strategy was used for NP surgery. If a patient had NP surgery before EOT/IPD CT scan, the data was censored after the time of the first NP surgery and the worst possible value (WP) was imputed in its place.
Time Frame: Baseline to EOT/IPD, up to 56 weeks
Population: CT analysis set and patients with a baseline CT who are rescued by SCS_NP by week 56
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 81 | 84
Score on a scale | -0.93 (5.06) | -0.20 (4.20)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; This endpoint compared the changes from baseline LMS score of benralizumab with placebo. H0: The change from baseline in LMS score is similar between benralizumab and placebo. H1: The change from baseline in LMS score is different between benralizumab and placebo; Test type: Superiority; p = 0.2375, ANCOVA — [p-value comment as in outcome 5, analysis 1]; ANCOVA following WP (WP for NP surgery), adjusting for treatment, baseline score, region (US/Non-US) and baseline comorbid asthma status; Mean Difference (Net) = -0.856, 95% CI 2-sided [-2.281 to 0.570]

12. Secondary Outcome: Percentage of Subjects With NP Surgery
Description: The percentage of patients who had nasal polyposis (NP) surgery or systemic corticosteroids use for nasal polyposis (SCS_NP) surgery up to week 56 was summarized and analyzed using the Cochran-Mantel-Haenszel test stratified by region (US vs non-US) and baseline comorbid asthma status (yes vs no).
Time Frame: Baseline to week 56
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 207 | 203
Participants | 33 | 37
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; This endpoint compared the proportion of subjects with NP surgery between benralizumab and placebo. H0: The proportion is similar between benralizumab and placebo. H1: The proportion is different between benralizumab and placebo; Test type: Superiority; p = 0.5419, Cochran-Mantel-Haenszel — This endpoint was not a part of the pre-specified testing strategy and was not tested for statistical significance. The p-value was considered nominal; The odds ratio estimate was obtained from the Cochran-Mantel-Haenszel test controlling for region (US/non-US) and baseline comorbid asthma status; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.51 to 1.43]

13. Secondary Outcome: Percentage of Subjects With SCS_NP
Description: The percentage of patients who had systemic corticosteroids (SCS) use for nasal polyposis (NP) surgery up to week 56 was summarized and analyzed using the Cochran-Mantel-Haenszel test stratified by region (US vs non-US) and baseline comorbid asthma status (yes vs no).
Time Frame: Baseline to week 56
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 207 | 203
Participants | 52 | 66
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; This endpoint compared the proportion of subjects with SCS_NP between benralizumab and placebo. H0: The proportion is similar between benralizumab and placebo. H1: The proportion is different between benralizumab and placebo; Test type: Superiority; p = 0.0913, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 12, analysis 1]; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.44 to 1.06]

14. Secondary Outcome: Percentage of Subjects With NP Surgery or SCS_NP
Description: as for outcome 12
Time Frame: Baseline to week 56
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 207 | 203
Participants | 72 | 91
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; This endpoint compared the proportion of subjects with NP surgery or SCS_NP between benralizumab and placebo. H0: The proportion is similar between benralizumab and placebo. H1: The proportion is different between benralizumab and placebo; Test type: Superiority; p = 0.0362, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 12, analysis 1]; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.44 to 0.97]

15. Secondary Outcome: Time to First SCS_NP up to Week 56
Description: The cumulative percentage and the corresponding 95% CI are based on the Kaplan-Meier estimates. Patients can have more than 1 rescue category during the study, and the first rescue per patient is considered. The time to first systemic corticosteroids for use for nasal polyposis (SCS_NP) up to week 56 was calculated based on the earliest occurrence of SCS_ NP and was calculated as follows: Time to first SCS_NP = Earlier of (Start date of first SCS use for NP) - date of randomization + 1. For patients who did not experience any SCS use for NP, the time to event was censored at earlier of (date of their week 56 visit, date of discontinuation). The time to first SCS use for NP surgery was analyzed using a Cox proportional hazard model with treatment arm, region (US vs non-US) and baseline comorbid asthma status (yes vs no) as covariates. A hazard ratio less than 1 indicates a lower rate of incidence for subjects on benra.
Time Frame: Baseline to week 56
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 207 | 203
months | 25.7 [20.2 to 32.3] | 33.5 [27.3 to 40.7]
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; The endpoint compared the rate of incidence of SCS_NP use between benralizumab and placebo. H0: The rate is similar between benralizumab and placebo. H1: the rate is different between benralizumab and placebo. Hazard ratio (HR) is benralizumab vs placebo and HR less than 1 indicates longer time to event; Test type: Superiority; p = 0.1505, Regression, Cox — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.53 to 1.10]

16. Secondary Outcome: Total Number of Courses of SCS for NP
Description: The total number of courses of systemic corticosteroids (SCS) use for nasal polyposis (NP) was summarized using descriptive statistics.
Time Frame: Baseline to week 56
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: number of courses
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 207 | 203
number of courses | 1.7 (0.93) | 1.6 (0.89)

17. Secondary Outcome: Total SCS_NP Dose (a) Used (mg)
Description: The total systemic corticosteroids (SCS) for nasal polyposis (NP) dose used (mg) was summarized using descriptive statistics.
Time Frame: Baseline to week 56
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 207 | 203
milligrams | 1083.2 (4044.29) | 435.2 (441.57)

18. Secondary Outcome: Total Duration of SCS_NP (Days)
Description: The total duration of systemic corticosteroids (SCS) for nasal polyposis (NP) in days was summarized using descriptive statistics.
Time Frame: Baseline to week 56
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 207 | 203
days | 17.6 (12.45) | 20.1 (34.68)

19. Secondary Outcome: Annual SCS_NP Use Rate Comparison by Period, Negative Binomial Model
Description: Annual systemic corticosteroids for nasal polyposis (SCS_NP) use rate =365.25×total number of courses of SCS_NP /total duration of follow-up within the treatment group (days). The estimated annual event rates, absolute differences, rate ratio and the corresponding confidence interval were based on a negative binomial model including covariates treatment group, region (US/non-US) and prior use of SCS_NP with total number of courses of SCS_NP as the outcome and the log of each subject's corresponding follow-up time up to week 56 as an offset variable in the model to adjust for subject's having different exposure times during which the events occur.
Time Frame: Baseline to week 56
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: number of courses for each patient
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 207 | 203
number of courses for each patient | 0.40 [0.30 to 0.52] | 0.50 [0.38 to 0.65]
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; The endpoint compared the rate of SCS_NP use between benralizumab and placebo. H0: The rate is similar between benralizumab and placebo. H1: the rate is different between benralizumab and placebo. Rate ratio is benralizumab vs placebo and Rate ratio less than 1 indicates less likely of SCS_NP use; Test type: Superiority; p = 0.2189, Negative Bionomial Model — [p-value comment as in outcome 12, analysis 1]; Model included treatment, US/non-US and prior use of SCS_NP with total number of courses of SCS_NP as outcome and log of follow-up time as an offset; Rate Ratio = 0.79, 95% CI 2-sided [0.54 to 1.15]

20. Secondary Outcome: Change From Baseline in TSS at Week 40
Description: Change from baseline in total symptom score (TSS) at week 40 was defined as the endpoint at week 40 minus baseline value. The TSS is defined as sum of first 8 NPSD components. Severity of each nasal symptoms over the past 24 hours is rated using response options: 0-none; 1-mild; 2-moderate; 3-severe. The TSS and the change from baseline were summarized every two weeks (bi-weekly). Baseline was the average of daily TSS responses from Day -13 to Day 1. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for nasal polyposis (SCS_NP) were set to missing. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied. In ANCOVA, a hybrid method of the WP after NP surgery, WOCF after SCS_NP and multiple imputation (MI) assuming MAR were used to build the complete imputation datasets for the analysis.
Time Frame: Baseline to week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 181
Score on a scale | -3.20 (6.90) | -1.38 (6.29)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; This endpoint compared the changes from baseline score between benralizumab and placebo. H0: The change from baseline score is similar between benralizumab and placebo. H1: The change from baseline score is different between benralizumab and placebo; Test type: Superiority; p = 0.0036, ANCOVA — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 1, analysis 1]; Median Difference (Net) = -1.854, 95% CI 2-sided [-3.101 to -0.608]

21. Secondary Outcome: Change From Baseline in Difficulty With Sleeping Due to Nasal Symptoms at Week 40
Description: Change from baseline in difficulty with sleeping due to nasal symptoms score at week 40 was defined as the endpoint at week 40 minus baseline value. The score was captured by an item in NPSD. The severity of difficulty with sleeping due to nasal symptoms over past 24 hours was rated using options: 0-none; 1-mild; 2-moderate; 3-severe. The score and change from baseline were summarized every two weeks (bi-weekly). Baseline was the average of daily responses from Day -13 to Day 1. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for nasal polyposis (SCS_NP) were set to missing. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied. In ANCOVA, a hybrid method of the WP after NP surgery, WOCF after SCS_NP and multiple imputation (MI) assuming missing at random were used to build the complete imputation datasets for the analysis
Time Frame: Baseline to week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 181
Score on a scale | -0.39 (1.06) | -0.19 (1.03)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.0941, ANCOVA — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.166, 95% CI 2-sided [-0.360 to 0.028]

22. Secondary Outcome: Change From Baseline in Difficulty With Daily Activities Due to Nasal Symptoms at Week 40
Description: Change from baseline in difficulty with daily activities due to nasal symptoms score at week 40 was defined as the endpoint at week 40 minus baseline value. The score was captured by an item in NPSD. The severity of difficulty with daily activities due to nasal symptoms over the past 24 hours was rated using options: 0-none; 1-mild; 2-moderate; 3-severe. The score and change from baseline were summarized every two weeks (bi-weekly). Baseline was average of daily responses from Day -13 to Day 1. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for nasal polyposis (SCS_NP) were set to missing. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied. In ANCOVA, a hybrid method of the WP after NP surgery, WOCF after SCS_NP and multiple imputation (MI) assuming MAR were used to build the complete imputation datasets for the analysis.
Time Frame: Baseline to week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 181
Score on a scale | -0.35 (1.04) | -0.11 (0.99)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.0246, ANCOVA — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.213, 95% CI 2-sided [-0.399 to -0.027]

23. Secondary Outcome: Change From Baseline in UPSIT Score in Males at Week 40
Description: Change from baseline in University of Pennsylvania Smell Identification Test (UPSIT) score at week 40 was defined as the endpoint value at week 40 minus the baseline value. The UPSIT is quantitative test of olfactory function. Scores were based on number of correctly identified odors (score range 0 to 40). Baseline was the last valid value on or prior to the date of randomization. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for nasal polyposis (SCS_NP) were set to missing. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied. In ANCOVA, a hybrid method of the WP after NP surgery, WOCF after SCS_NP and multiple imputation (MI) assuming missing at random were used to build the complete imputation datasets for the analysis.
Time Frame: Baseline to week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 109 | 89
Score on a scale | -0.20 (10.29) | 0.09 (8.05)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.5833, ANCOVA — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.672, 95% CI 2-sided [-1.730 to 3.074]

24. Secondary Outcome: Change From Baseline in UPSIT Score in Females at Week 40
Description: Change from baseline in University of Pennsylvania Smell Identification Test (UPSIT) score at week 40 was defined as the endpoint value at week 40 minus the baseline value. The UPSIT is quantitative test of olfactory function. Scores are based on number of correctly identified odors (score range 0 to 40). Baseline was the last valid value on or prior to the date of randomization. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for nasal polyposis (SCS_NP) were set to missing. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied. In ANCOVA, a hybrid method of the WP after NP surgery, WOCF after SCS_NP and multiple imputation (MI) assuming missing at random were used to build the complete imputation datasets for the analysis.
Time Frame: Baseline to week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 53 | 74
Score on a scale | 1.66 (8.86) | -1.32 (7.66)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.0619, ANCOVA — [p-value comment as in outcome 12, analysis 1]; [statistical method as in outcome 1, analysis 1]; Median Difference (Net) = 2.684, 95% CI 2-sided [-0.134 to 5.502]

25. Secondary Outcome: Change From Baseline in Sinus Severity Score at EOT/IPD
Description: Change from baseline in sinus severity score at end of treatment (EOT)/investigational product discontinuation (IPD) was defined as the endpoint value at EOT/IPD minus the baseline value. Quantitative assessment of sinus CT image data was used to derive an objective measure of sinus disease burden called sinus severity score. The sinus severity score is defined as (sinus mucosal volume)/(sinus mucosal volume + sinus air volume)×100. A composite strategy was used for NP surgery. If a patient had NP surgery before EOT/IPD CT scan, the data was censored after the time of the first NP surgery and the worst possible value (WP) was imputed in its place. In calculation of summary statistics (mean and standard deviation), the WP for NP surgery rescued subjects was applied. In ANCOVA, following WP (WP for NP surgery rescued subjects), model included treatment, baseline score, region (US/Non-US) and baseline comorbid asthma status.
Time Frame: Baseline to EOT/IPD, up to 56 weeks
Population: CT analysis set and patients with a baseline CT who are rescued by SCS_NP by week 56. Patients who had not been rescued and whose post-baseline observation was missing at the timepoint of interest are excluded from this analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 86 | 84
Score on a scale | -3.48 (24.24) | 0.79 (17.29)
Statistical Analysis 1: Comparison: Benra 30 mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.1020, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Following WP (WP for NP surgery rescued subjects), model included treatment, baseline score, region (US/Non-US) and baseline comorbid asthma status; Median Difference (Net) = -5.057, 95% CI 2-sided [-11.129 to 1.015]

26. Secondary Outcome: Change From Baseline in SF-36v2 Physical Component Summary at Week 56
Description: Change from baseline in SF-36v2 physical component summary (PCS) at week 56 was defined as the endpoint value at week 56 minus the baseline value. The Short Form 36-item Health survey (SF-36v2) is a 36-item, self-report survey of functional health and wellbeing, with 4-week recall period. Responses to SF-36v2 were used to compute an 8-domain profile of functional health and well-being scores. PCS score is computed from 8 subscale scores to give a broader metric of physical health-related quality of life. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. Non-rescued patients whose post-baseline observations were all missing were excluded from this analysis. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 185
Score on a scale | -1.557 (17.7075) | -3.185 (17.4189)

27. Secondary Outcome: Change From Baseline in SF-36v2 Mental Component Summary at Week 56
Description: Change from baseline in SF-36v2 mental component summary (MCS) at week 56 was defined as the endpoint value at week 56 minus the baseline value. The Short Form 36-item Health survey (SF-36v2) is a 36-item, self-report survey of functional health and wellbeing, with 4-week recall period. Responses to SF-36v2 were used to compute an 8-domain profile of functional health and well-being scores. MCS score is computed from 8 subscale scores to give a broader metric of mental health-related quality of life. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. Non-rescued patients whose post-baseline observations were all missing were excluded from this analysis. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 185
Score on a scale | -2.263 (18.4094) | -4.182 (19.3697)

28. Secondary Outcome: Change From Baseline in SF-36v2 Physical Functioning at Week 56
Description: Change from baseline in SF-36v2 physical functioning score at week 56 was defined as the endpoint value at week 56 minus the baseline value. The Short Form 36-item Health survey (SF-36v2) is a 36-item, self-report survey of functional health and wellbeing, with 4-week recall period. Responses to SF-36v2 were used to compute an 8-domain profile of functional health and well-being scores. Physical functioning is one of the 8-domain profile. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. Non-rescued patients whose post-baseline observations were all missing were excluded from this analysis. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 185
Score on a scale | 0.080 (14.8681) | -0.911 (14.6581)

29. Secondary Outcome: Change From Baseline in SF-36v2 Role Limitations Due to Physical Health at Week 56
Description: Change from baseline in SF-36v2 role limitations due to physical health score at week 56 was defined as the endpoint value at week 56 minus the baseline value. The Short Form 36-item Health survey (SF-36v2) is a 36-item, self-report survey of functional health and wellbeing, with 4-week recall period. Responses to SF-36v2 were used to compute an 8-domain profile of functional health and well-being scores. Role limitations due to physical health is one of the 8-domain profile. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. Non-rescued patients whose post-baseline observations were all missing were excluded from this analysis. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 185
Score on a scale | 1.576 (13.4610) | 0.025 (13.3886)

30. Secondary Outcome: Change From Baseline in SF-36v2 Bodily Pain at Week 56
Description: Change from baseline in SF-36v2 bodily pain score at week 56 was defined as the endpoint value at week 56 minus the baseline value. The Short Form 36-item Health survey (SF-36v2) is a 36-item, self-report survey of functional health and wellbeing, with 4-week recall period. Responses to SF-36v2 were used to compute an 8-domain profile of functional health and well-being scores. Bodily pain is one of the 8-domain profile. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. Non-rescued patients whose post-baseline observations were all missing were excluded from this analysis. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 185
Score on a scale | 0.982 (15.0935) | -1.066 (15.3689)

31. Secondary Outcome: Change From Baseline in SF-36v2 General Health Perceptions at Week 56
Description: Change from baseline in SF-36v2 general health perceptions score at week 56 was defined as the endpoint value at week 56 minus the baseline value. The Short Form 36-item Health survey (SF-36v2) is a 36-item, self-report survey of functional health and wellbeing, with 4-week recall period. Responses to SF-36v2 were used to compute an 8-domain profile of functional health and well-being scores. General health perceptions is one of the 8-domain profile. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. Non-rescued patients whose post-baseline observations were all missing are excluded from this analysis. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 185
Score on a scale | 0.445 (14.2295) | -1.064 (13.6387)

32. Secondary Outcome: Change From Baseline in SF-36v2 Vitality at Week 56
Description: Change from baseline in SF-36v2 vitality score at week 56 was defined as the endpoint value at week 56 minus the baseline value. The Short Form 36-item Health survey (SF-36v2) is a 36-item, self-report survey of functional health and wellbeing, with 4-week recall period. Responses to SF-36v2 were used to compute an 8-domain profile of functional health and well-being scores. Vitality is one of the 8-domain profile. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. Non-rescued patients whose post-baseline observations were all missing were excluded from this analysis. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 185
Score on a scale | 1.913 (12.9999) | -0.594 (13.5861)

33. Secondary Outcome: Change From Baseline in SF-36v2 Social Functioning at Week 56
Description: Change from baseline in SF-36v2 social functioning score at week 56 was defined as the endpoint value at week 56 minus the baseline value. The Short Form 36-item Health survey (SF-36v2) is a 36-item, self-report survey of functional health and wellbeing, with 4-week recall period. Responses to SF-36v2 are used to compute an 8-domain profile of functional health and well-being scores. Social functioning is one of the 8-domain profile. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. Non-rescued patients whose post-baseline observations were all missing were excluded from this analysis. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 185
Score on a scale | 0.262 (15.1786) | -1.247 (15.9512)

34. Secondary Outcome: Change From Baseline in SF-36v2 Role Limitations Due to Emotional Problems at Week 56
Description: Change from baseline in SF-36v2 role limitations due to emotional problems score at week 56 was defined as the endpoint value at week 56 minus the baseline value. The Short Form 36-item Health survey (SF-36v2) is a 36-item, self-report survey of functional health and wellbeing, with 4-week recall period. Responses to SF-36v2 were used to compute an 8-domain profile of functional health and well-being scores. Role limitations due to emotional problems is one of the 8-domain profile. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. Non-rescued patients whose post-baseline observations were all missing were excluded from this analysis. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 185
Score on a scale | -0.492 (17.1261) | -1.825 (16.6618)

35. Secondary Outcome: Change From Baseline in SF-36v2 Mental Health at Week 56
Description: Change from baseline in SF-36v2 mental health score at week 56 was defined as the endpoint value at week 56 minus the baseline value. The Short Form 36-item Health survey (SF-36v2) is a 36-item, self-report survey of functional health and wellbeing, with 4-week recall period. Responses to SF-36v2 were used to compute an 8-domain profile of functional health and well-being scores. Mental health is one of the 8-domain profile. Data collected after nasal polyposis (NP) surgery and/or systemic corticosteroids for NP (SCS_NP) were set to missing. Non-rescued patients whose post-baseline observations were all missing were excluded from this analysis. In calculation of summary statistics (mean and standard deviation), the worst-possible (WP) after NP surgery and worst-observation carried forward (WOCF) after SCS_NP were applied.
Time Frame: Baseline to week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benra 30 mg | Placebo
Number analyzed (Participants) | 191 | 185
Score on a scale | -1.506 (16.5930) | -3.308 (17.2382)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until end of study, up to 603 days.
Description: For analysis of Adverse Events Safety analysis set is used. Safety analysis set : All randomized participants who received at least one dose of study drug.
Arm/Group | Benra 30 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/207 | 0/203
Serious Adverse Events (participants affected / at risk) | 25/207 | 19/203
Other Adverse Events (participants affected / at risk) | 64/207 | 83/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg (N=207) | Placebo (N=203)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 2 (3) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mucoepidermoid carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrospinal fistula (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg (N=207) | Placebo (N=203)
Nasopharyngitis (Infections and infestations) | 37 (57) | 43 (54)
Viral upper respiratory tract infection (Infections and infestations) | 7 (9) | 14 (15)
Headache (Nervous system disorders) | 7 (9) | 16 (18)
Asthma (Respiratory, thoracic and mediastinal disorders) | 21 (30) | 30 (54)

LIMITATIONS AND CAVEATS:
During COVID-19 pandemic, for ongoing patients, patient dosing, scheduled visits, and nasal endoscopies are inevitable impacted. Week 40 was made as the primary timepoint to mitigate the impact of COVID disruptions on the primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT03401229/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT03401229/SAP_001.pdf